CLINICAL TRIAL: NCT00907205
Title: A Phase I Open Label Safety, Pharmacokinetic and Pharmacodynamic Dose Escalation Study of SF1126, A PI3 Kinase (PI3K) Inhibitor, Given Twice Weekly By IV Infusion To Patients With Advanced or Metastatic Tumors
Brief Title: A Dose Escalation Study of SF1126, a PI3 Kinase (PI3K) Inhibitor, Given By Intravenous (IV) Infusion in Patients With Solid Tumors
Acronym: SF112600106
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Semafore Pharmaceuticals (Industry)
Collaborators: SignalRX Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF1126-001-06
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Advanced or Metastatic Solid Tumors; Cancer; Solid Cancers
Keywords: Advanced Solid Tumors; Metastatic Solid Tumors; PI3K; PI3K Inhibitors; PI3 Kinase Inhibitors; mTORC inhibitor; mTORC1 inhibitor; mTORC2 inhibitor; vascular targeted; conjugate
MeSH Terms: conditions — Neoplasms | interventions — SF 1126

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SF1126 (Experimental): Twice weekly IV infusion
  Interventions: Drug: SF1126

INTERVENTIONS:
Drug: SF1126 — Dose Escalating with 3+ patients in each cohort

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SF1126 in patients with advanced or metastatic tumors by assessing the dose limiting toxicities (DLTs) and defining the maximum tolerated dose given twice per week for 4 weeks and ultimately define a recommended phase II dose.

DETAILED DESCRIPTION:
SF1126 is a conjugate containing a vascular targeted pan-PI3K inhibitor that selectively inhibits all PI3K class I isoforms and other key members of the PI3K superfamily, including mTORC1/2, DNA-PK, PLK-1, CK2, ATM and PIM-1. SF1126 is designed to inhibit both angiogenesis and cell proliferation by targeting and binding to specific integrins such as αγβ3 that are expressed on the surface of new tumor vasculature and within the tumor compartment. In preclinical xenograft models SF1126 has demonstrated broad activity as a single agent; synergy with commonly used chemotherapy agents, targeted agents, and radiation; and has been shown to reverse resistance mediated through the PI3K/PTEN pathway.

ELIGIBILITY:
Inclusion Criteria:

To qualify for enrollment, all of the following criteria must be met:

* Written informed consent.
* At least 18 years old.
* Accrual will be limited to patients with tumor types that in the opinion of the investigator is known to have PTEN loss or PI3 Kinase mutations potentially important in the biology of their cancer.
* Only patients with histologically confirmation of advanced solid malignant tumor which is refractory to standard therapies or which no standard therapy exists.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Life expectancy of > or = 12 weeks.
* Female subjects are eligible to enter and participate in the study if: they are non-childbearing potential, had a hysterectomy, had a bilateral oophorectomy (ovariectomy), had a bilateral tubal ligation, post-menopausal or childbearing potential with a negative serum pregnancy test at screening and agrees to protection by IUD, vasectomized partner, complete abstinence, double barrier contraception.
* male patients with childbearing potential must agree to use adequate contraception while on study.
* patients on active therapy with well-controlled diabetes as defined by fasting glucose < 160mg/dL.

Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before entry, and stable without steroid treatment for at least 4 weeks.
* Inadequate bone marrow reserve as demonstrated by an absolute neutrophil count <1.5 x 10^9/L or platelet count < 100 x 10^9/L (can not be post-transfusion) or hemoglobin <9 g/dL (can be post-transfusion).
* Serum bilirubin > or = 1.2 times the upper limit of normal.
* An ALT or AST level > or = 2.5 times the upper limit of normal. If documented liver metastases are present, the ALT or AST levels must still be less than 2.5 times the upper limit of normal.
* Serum creatinine > 1.5 times the upper limit of normal or a creatinine clearance of < or = 50mL/min calculated by the Cockcroft-Gault equation.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac [including life threatening arrhythmias], hepatic, or renal disease.
* Unresolved toxicity ≥CTC Grade 2 from previous anti-cancer therapy except alopecia (if applicable) unless agreed that the patient can be entered after discussion with the Medical Monitor.
* QTc prolongation defined as a QTc >450 ms for males or >470ms for females (Fridericia) for 3 consecutive ECGs; OR prior history of cardiovascular disease including heart failure that meets New York Hearth Association (NYHA) class III and IV definitions, OR history of myocardial infarction/active ischemic heart disease within one year of study entry; OR uncontrolled dysrhythmias; OR poorly controlled angina.
* Participation in a trial of an investigational agent within the prior 30 days.
* Pregnant or breast-feeding females.
* High volume peritoneal or pleural effusions requiring a tap more frequently than every 14 days.
* History of other malignancies except curatively excised carcinoma in situ of the cervix, non-melanomatous skin carcinoma or superficial bladder cancer or other solid tumors curatively treated with no evidence of disease for > or = 5 years. Other cases will be reviewed and possibly allowed if discussed with and approved by Medical Monitor.
* Patients receiving therapeutic doses of Warfarin.
* Any concurrent condition which in the investigator's opinion makes it undesirable for the subject to participate in this trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the dose limiting toxicities (DLTs) of SF1126 and the maximum tolerated dose given twice per week for 4 weeks and ultimately define a recommended phase II dose. | Assessed at each visit and end of cycle 1

SECONDARY OUTCOMES:
To assess any preliminary evidence of anti-tumor activity observed with SF1126 | Through study completion or early study discontinuation
To characterize the pharmacokinetics following the IV doses on Days 1 and 28 | Cycle 1 Days 1 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Durden, MD, PhD, Study Chair — SignalRX Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Scottsdale Clinical Research Institute, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

REFERENCES:
- [Result] Mahadevan D, Chiorean EG, Harris WB, Von Hoff DD, Stejskal-Barnett A, Qi W, Anthony SP, Younger AE, Rensvold DM, Cordova F, Shelton CF, Becker MD, Garlich JR, Durden DL, Ramanathan RK. Phase I pharmacokinetic and pharmacodynamic study of the pan-PI3K/mTORC vascular targeted pro-drug SF1126 in patients with advanced solid tumours and B-cell malignancies. Eur J Cancer. 2012 Dec;48(18):3319-27. doi: 10.1016/j.ejca.2012.06.027. Epub 2012 Aug 23. PMID 22921184
- See also: SignalRx Pharmaceuticals Website — http://www.signalrx.com